CLINICAL TRIAL: NCT02464254
Title: Intervention to Support Participation in Regular Exercise in the Elderly (INSPIRE)
Acronym: INSPIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1303013686; 1K23AG042869-01A1 (NIH)
Record Dates: First submitted 2015-06-02; First posted 2015-06-08 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Chronic Illnesses
Keywords: Physical activity, positive affect, older adults, aging
MeSH Terms: conditions — Chronic Disease; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity plus positive affect (Experimental): Subjects will be randomized to a physical activity goal and the positive affect component
  Interventions: Behavioral: Physical activity plus positive affect; Behavioral: Physical activity plus education
- Physical activity plus education (Active Comparator): Subjects will be randomized to a physical activity goal and education
  Interventions: Behavioral: Physical activity plus education

INTERVENTIONS:
Behavioral: Physical activity plus positive affect — Subjects will be randomized to a physical activity goal and will receive the positive affect component.
  Arms: Physical activity plus positive affect
Behavioral: Physical activity plus education — Subjects will be randomized to a physical activity goal and will receive the educational component.

SUMMARY:
The investigators will conduct a 1-year prospective and randomized study to evaluate the initial efficacy of positive affect vs. an educational control to motivate physical activity in older adults with high burdens of chronic disease.

DETAILED DESCRIPTION:
Older adults with multiple chronic diseases are at high risk for both disability and adverse clinical events, outcomes that can be improved with physical activity, but there have been no trials to establish physical activity recommendations or clinical guidelines for this vulnerable population. A recent randomized controlled trial conducted by Dr. Peterson established the efficacy of inducing positive affect-a feeling of happiness and well-being-in motivating physical activity in older adults with cardiovascular disease. This new randomized controlled trial will pilot test the a new PAIRE (Positive Affect Induction for Regular Exercise) intervention that is specific to older adults with multiple high-risk chronic illnesses versus an educational control group. This work is innovative because it will translate the benefits of a proven intervention focused on positive affect to increase physical activity in older adults with multiple high-risk chronic illnesses, one that is tailored to the clinical and psychosocial challenges of this particularly vulnerable population. This work is significant because an effective intervention promoting physical activity will improve outcomes for older adults with multiple high-risk chronic diseases, and currently one does not exist.

ELIGIBILITY:
Inclusion Criteria:

* Charlson Index greater or equal to 3

Exclusion Criteria:

1. Cognitive impairment
2. Inability to walk
3. < 12 month anticipated survival
4. enrollment in other behavioral programs
5. lack of medical approval to participate
6. substance/alcohol dependence or participation in a substance abuse treatment program within 12 months
7. major psychiatric illness.

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Kilocalories/week assessed by Objective measure of activity with accelerometry | baseline to 12 months
  FitBit

SECONDARY OUTCOMES:
Kilocalories/week assessed by Subjective measure of activity by self-report | baseline to 12 months
Function/disability assessed by objective and subjective reports of functional ability | baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Janey Peterson, EdD MS RN, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the main article reporting the results, after deidentification
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal